CLINICAL TRIAL: NCT01896739
Title: A Multicentre, Comparative, Open-label, Randomized, Phase III Study to Assess the Immunogenicity and Safety of EutravacTMinj (DTaP-HB Combined Vaccine) Administered at 2,4, 6 Months of Age Compared With DTaP Vaccine at 2, 4, 6 Months of Age Combined Administered Monovalent Hepatitis B Vaccine Administered at Birth, 1, 6 Months of Age in Healthy Infants.
Brief Title: A Phase III Study to Assess the Immunogenicity and Safety of Eutravac (DTap-HB Combined Vaccine) With DTaP and Hepatitis B Vaccines in Healthy Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LG-VACL004
Record Dates: First submitted 2013-07-08; First posted 2013-07-11 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Healthy Infants
Keywords: Healthy infants with over than 37 weeks gestation periods.; over than 2.5Kg at at birth weight.
MeSH Terms: interventions — Euvax-B; Hepatitis B Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Experimental group with 0-2-4-6 schedule (Experimental): HB at 0, Eutravac at 2-4-6
  Interventions: Biological: Eutravac
- Active comparator group with 0-2-4-6 schedule (Active Comparator): Separate injection of DTaP and HB at 2-4-6 (for DTaP) and 0-1-6 (HB)
  Interventions: Biological: Eutravac
- Experimental group with 2-4-6 schedule (Experimental): Eutravac at 2-4-6
  Interventions: Biological: Eutravac
- Active comparator group with 2-4-6 schedule (Active Comparator): Separate injection of DTaP and HB at 2-4-6 (for DTaP) and 0-1-6 (HB)
  Interventions: Biological: Eutravac

INTERVENTIONS:
Biological: Eutravac
  Other Names: LG DTaP Vaccine Inj. (DTaP); Euvax B (Hepatitis B); Hepavax (Hepatitis B)

SUMMARY:
To evaluate and compare the immunogenicity of Eutravac (Diphtheria-Tetanus-acellular Pertussis [DTaP] Hepatitis B [HB] combined) vaccine with separate but simultaneous administrations of DTaP and HB vaccine each administered to healthy infants, as measured by seroprotection/vaccine response rates 4-8 weeks post-final immunisation.

ELIGIBILITY:
Inclusion Criteria:

* Were healthy, male or female infants born at full term pregnancy (≥37 weeks) with a birth weight ≥2.5 kg to mothers with a negative HBsAg serology, documented prior to giving birth as per routine, site-specific ante-natal care procedures.
* Signed parental or legally acceptable representative's informed consent was obtained

Exclusion Criteria:

* Evidence of an acute febrile illness with axillary temperature ≥37.5℃ on the day of the vaccination. Infants with symptoms of minor illness eg, mild gastroenteritis, mild upper respiratory tract infection and who did not have a temperature ≥37.5℃ on the day of the vaccination could be included at the Investigator's discretion
* History of diphtheria, tetanus, pertussis or hepatitis B disease
* History of any vaccine-related hypersensitivity or anaphylactic reaction after previous administration of Euvax B

Max Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 289 (Actual)
Dates: Start 2009-08; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Seroprotection rate | After final immunisation at 4-8 weeks

CONTACTS AND LOCATIONS:
Locations (7):
- South Korea (7):
  - Daejeon St. Mary's Hospital, Daejeon, Daejeon
  - The Catholic University of Korea ST. Vincent's Hospital, Suwon, Gyeonggi-do
  - Inha University Hospital, Incheon, Incheon
  - Jeju National University Hospital, Jeju City, Jeju-do
  - Kyung Hee University Hospital, Seoul, Seoul
  - Cha Hospital, Seoul, Seoul
  - Korea Cancer Center Hospital, Seoul, Seoul